CLINICAL TRIAL: NCT01510873
Title: Health-related Quality of Life and Fatigue in Adult Patients With Primary Immune Thrombocytopenic Purpura (pITP).
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: QoL-ITP0411
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: Health-related quality of life; Fatigue; pITO; Primary Immune Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Newly Diagnosed pITP: Patients within 3 months from diagnosis.
  Interventions: Other: HRQOL evaluation
- Persistent pITP: Patients between 3 to 12 months from diagnosis; includes patients not reaching spontaneous remission or not maintaining complete response off therapy.
  Interventions: Other: HRQOL evaluation
- Chronic pITP: Patients with ITP lasting for more than 12 months.
  Interventions: Other: HRQOL evaluation

INTERVENTIONS:
Other: HRQOL evaluation — Patients will be asked to complete a Questionnaire (i.e. HRQOL Survey Packet) that will cover a number of issues. These will include socio-demographic aspects, HRQOL information, symptom burden, clinical decision-making, social support and psychological wellbeing. Most of these information will be collected through well known psychometrically sound questionnaires. The copyright for using standardized questionnaires will be obtained, from the appropriate copyright holders, for the purpose of this research.
  The Questionnaire properly formatted will be distributed to all participating Centers prior to study start.

SUMMARY:
Symptoms of Primary Immune Thrombocytopenic Purpura (pITP), such as spontaneous bruising, menorrhagia, mucosal bleeding and other symptoms might significantly affect the HRQOL of pITP patients. However, very little evidence exists on HRQOL outcomes in patients diagnosed with pITP. The investigators project will aim at providing scientific community solid evidence based data on the extent to which HRQOL is compromised and in which specific area.

The purpose of this study is thus to compare generic Health-related Quality of Life (HRQOL) profiles of adult patients with primary Immune Thrombocytopenic Purpura (pITP) with that of a matched Italian population control Group.

DETAILED DESCRIPTION:
OBJECTIVES:

The primary objective is to compare HRQOL of patients with pITP with that of a matched Italian population control Group.

Secondary objectives include evaluation of:

* Patient-reported fatigue amongst the three different pITP groups.
* Social support and psychological wellbeing as a possible determinant of HRQOL.
* Possible association between socio-demographic (e.g., age, living arrangements, education and employment status) and clinical variables (e.g., time from diagnosis, and current treatment if any) with patient reported health outcomes (e.g., HRQOL, fatigue, and social support).
* To assess patients' preferences for involvement in treatment decision-making and the relationships between preferences and patient characteristics and to compare patient's stated preferences for involvement in treatment decision with the perceptions of their treating physicians (only for Newly Diagnosed pITP).

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of pITP in any phase of the disease;
* Patients aged at least 18 years;
* Informed consent provided

Exclusion Criteria:

* Participating in other HRQOL investigations that might interfere with this study
* Having any psychiatric condition or major cognitive impairment hampering self-reported HRQOL evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 years of age or older) with confirmed diagnosis of pITP in any phase of the disease
Sampling Method: Non-Probability Sample
Enrollment: 424 (Actual)
Dates: Start 2011-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Comparison of HRQOL of patients with pITP with that of a matched Italian population control Group. | By the end of the study.

SECONDARY OUTCOMES:
Patient-reported fatigue amongst the three different pITP groups | By the end of the study.
Patient-reported fatigue amongst the three different pITP groups. | By the end of the study.
Possible association between socio-demographic and clinical variables with patient reported health outcomes. | By the end of the study.
To assess patients' preferences for involvement in treatment decision-making. | By the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Efficace, PhD, Principal Investigator — GIMEMA DATA CENTER, ROME, ITALY
Locations (29):
- Italy (29):
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Ospedale Generale Regionale "F. Miulli", Acquaviva delle Fonti
  - Azienda Ospedaliero-Universitaria Policlinico Consorziale, Bari
  - Azienda Sanitaria Locale BA - Ospedale di Venere, Bari
  - Ospedali Riuniti di Bergamo, Bergamo
  - Ospedale Binaghi, Cagliari
  - Ospedale Businco, Cagliari
  - U.O.C. di Onco-Ematologia - Centro di Ricerca e Formazione ad Alta tecnologia nelle Scienze Biomediche, Campobasso
  - US Dipartimentale - Centro per le malattie del sangue - Ospedale Civile - S.Giacomo, Castelfranco Veneto
  - Azienda Ospedaliero Universitaria, Foggia
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - DIMI- Clinica Ematologica - Università degli studi di Genova, Genova
  - Ospedale Santa Maria Goretti, Latina
  - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte", Messina
  - Azienda Ospedaliera Universitaria - Policlinico "G. Martino", Messina
  - Azienda Ospedaliero - Universitaria di Modena, Modena
  - Azienda Ospedaliera "S. Gerardo dei Tintori", Monza
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Ospedale S. Luigi Gonzaga, Orbassano
  - Azienda Ospedaliera Universitaria - Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliero - Universitaria di Parma, Parma
  - Azienda Ospedaliera "Bianchi - Melacrino - Morelli", Reggio Calabria
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - U.O.S.A. Ematologia ASL RMA Presidio Nuovo Regina Margherita, Roma
  - UOC Pronto Soccorso e Accettazione Ematologica - Dipartimento Biotecnologie Cellulari ed Ematologia - Università degli Studi di Roma "Sapienza", Rome
  - U.O. Ematologia, Azienda Ospedaliera Universitaria Senese, Siena
  - Azienda Ospedaliero - Universitaria "San Giovanni Battista", Torino
  - Azienda Ospedaliera, Treviglio
  - ULSS N.6 Ospedale San Bortolo, Vicenza

REFERENCES:
- See also: GIMEMA — http://www.gimema.it